CLINICAL TRIAL: NCT06430684
Title: Feasibility Trial of Sodium-GLucose CoTransporter 2 INhibitors in Pediatric Chronic KIDney DiSease
Acronym: SGLT2I-IN-KIDS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Alexander Kula, Assistant Professor of Pediatrics (Nephrology), Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGLT2I-IN-KIDS; K23DK138313 (NIH)
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Diseases; Pediatric Kidney Disease
Keywords: Sodium Glucose Co-Transporter 2 Inhibitor; SGLT2i; Pediatric CKD; Feasibility Study; Clinical Trial
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Empagliflozin 10mg daily for 3 months (n=20)
  Interventions: Drug: Empagliflozin 10 MG
- Standard of Care (No Intervention): Participants will not take empagliflozin (n=20)

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Empagliflozin is a sodium glucose co-transporter 2 inhibitor (SGLT2i) that is approved for the treatment of chronic kidney disease (CKD) in persons aged 18 years or older
  Arms: Treatment

SUMMARY:
The goal of this study is to learn if a clinical trial of sodium-glucose co-transporter 2 inhibitors (SGLT2i) is possible in youth with chronic kidney disease (CKD). The investigators also plan to explore whether treatment with SGLT2i (Empagliflozin) helps improve risk factors for worsening kidney and heart disease. The main questions are:

1. Is enrolling 40 youth with CKD into a clinical trial of empagliflozin feasible (ie achievable)?
2. Does taking empagliflozin for 3 months result in positive changes in blood, urine, and heart function tests?

Participants will be randomly selected (like flipping a coin) to either receive empagliflozin or not start treatment with empagliflozin and remain on their usual care.

Study Procedures Include

* For participants randomly selected for treatment, take empagliflozin once daily for 3 months
* Phone calls with researchers every 2 weeks for check-ins
* For participants taking empagliflozin, clinic visits 4 and 8 weeks after starting for check-ups and tests
* All study participants will have clinic visits at the beginning and end (3 months) where researchers will collect information about their health and perform tests

ELIGIBILITY:
Inclusion Criteria:

* Stage 3-4 CKD; estimated GFR using CKiD U25-creatinine equation 20-60mL/min/1.73m2

Exclusion Criteria:

* Heart Disease
* Diabetes
* Pregnancy
* Recipient of solid organ transplant
* history of chemotherapy or stem cell transplant
* moderate to severe persistent asthma
* liver disease
* class 2 or greater obesity
* inability to follow study procedures due to cognitive impairment
* obstructive uropathy or requirement for intermittent urinary catheterization
* systolic blood pressure <100mgHg
* orthostatic hypotension
* current use of an SGLT2i
* anticipated need for titration of anti-hypertensives within 3 months
* active use of any immunosuppressive medications
* lack of clearance by primary nephrologist for participation

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who complete all study procedures | 4 years
  Compared to the number recruited, how many participants complete the study

SECONDARY OUTCOMES:
Systolic Blood Pressure | 3 months
  In-clinic systolic blood pressure
Serum N-terminal pro-brain natruetic peptide (NT-proBNP) | 3 months
Urine Albumin to Creatinine Ratio (UACr) | 3 months
Left Atrial Reservoir Strain | 3 months
  Measuring using echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No